CLINICAL TRIAL: NCT04762147
Title: Comparison of Perioperative Analgesia Between Intravenous Paracetamol and Fentanyl for Rigid Hysteroscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dileep Kumar, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4370-Ane-ERC-16
Record Dates: First submitted 2021-02-02; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Analgesia; Effect of Drug
Keywords: ParacetamolGeneral anaesthesia; Fentanyl; General Anaesthesia; Hysterescopy
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol group-P (Experimental): Paracetamol 15mg/Kg was dministered 30 minutes before the start of surgery
  Interventions: Drug: paracetamol, the group P
- Fentanyl group-F (Active Comparator): Fentanyl 2mcg/kg was administered at the time induction of anaesthesia
  Interventions: Drug: fentanyl, group-F administered as an active comparator

INTERVENTIONS:
Drug: paracetamol, the group P — The paracetamol was administered 30 minutes before the start of surgery for intra-operative and post-operative analgesia in patients undergoing for hysteroscopy
  Arms: Paracetamol group-P
Drug: fentanyl, group-F administered as an active comparator — The fentanyl 2mcg/kg was administered at the time induction of anaesthesia for intra-operative and post-operative analgesia in patients undergoing for hysteroscopy
  Arms: Fentanyl group-F

SUMMARY:
Objective of study:

To compare the efficacy of intravenous paracetamol and fentanyl for intra-operative and post-operative pain relief in patients undergoing diagnostic and therapeutic hysteroscopy.

Hypothesis of study:

There is no difference in pain control between intravenous fentanyl and paracetamol in patients undergoing hysteroscopy.

DETAILED DESCRIPTION:
Intraoperative pain assessment will be based on:

Hemodynamic vital (SBP, DBP. MAP and HR) increase 20% from the baseline will be observed and assumed pain.

Postoperative pain assessment will be based on:

Mean Pain score :Visual analogue pain scale (VAS) of 0-10 cms will be used to assess the pain at the end of the procedure.

Diagnostic hysteroscopy:

Patients presenting with abnormal premenopausal or postmenopausal uterine bleeding, pain, infertility, intrauterine adhesions, endometrial biopsy, foreign body.

Therapeutic hysteroscopy:

To remove IUD, uterine polyps, fibroid, foreign body and submucosal fibroids, sterilization.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* American Society of Anaesthesiologists (ASA) grade I & II

Exclusion Criteria:

* Patients with anticipated difficult airway
* Gastro-oesophageal reflux disorder
* Body mass index (BMI) >30kg/m2
* Known Hepatic disorder
* Known ischemic heart disease
* History of hypersensitivity reactions to paracetamol and fentanyl or already taking paracetamol and fentanyl
* Patient experiencing the iatrogenic intra-operative uterine perforation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Hysteroscopy is procedure perfomed in females only
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Intra-operative pain assessment was based on the changes at each five minutes interval in systolic and diastolic blood pressure | Time frame was zero to 2 hours and data recordings were at 5 minutes interval from start from the surgical stimulation till the completion of the surgical procedure
  To assess the intra-operative pain by changes in hemodynamic parameters such as systolic blood pressure, diastolic blood pressure rising from the 20 percent of baseline value were considered that the patient is experiencing pain
Intra-operative pain assessment was based on changes in each five minutes interval in mean arterial blood pressure | Time frame was zero to 2 hours and data recordings were at 5 minutes interval from start from the surgical stimulation till the completion of the surgical procedure
  To assess the intra-operative pain by changes in hemodynamic parameters such as mean arterial blood pressure rising from the 20 percent of baseline value were considered that the patient is experiencing pain
Intra-operative pain assessment was based on changes in each five minutes interval in heart rate | Time frame was zero to 2 hours and data recordings were at 5 minutes interval from start from the surgical stimulation till the completion of the surgical procedure
  To assess the intra-operative pain by changes in hemodynamic parameters such as heart rate rising from the 20 percent of the baseline value were considered that the patient is experiencing pain
Post-operative pain assessed by using the visual analogue pain scale (VAS): Immediately after anaesthesia | Immediately post-anaesthesia
  To assess the postoperative pain by using the visual analogue pain scale (VAS) by using the scale in numbers from 0-10 cm in post anesthesia care unit.
  Note:
  Mild pain was considered score from 0 to 3, Moderate pain was labelled the score from 4 to 6 and Severe pain was considered the score from 7 to 10
Post-operative pain assessed by using the visual analogue pain scale (VAS): 15 minutes after anaesthesia | 15 minutes post-anaesthesia
  To assess the postoperative pain by using the visual analogue pain scale (VAS) by using the scale in numbers from 0-10 cm in post anesthesia care unit.
  Note:
  Mild pain was considered score from 0 to 3, Moderate pain was labelled the score from 4 to 6 and Severe pain was considered the score from 7 to 10
Post-operative pain assessed by using the visual analogue pain scale (VAS): 30 minutes after anaesthesia | 30 minutes post-anaesthesia
  To assess the postoperative pain by using the visual analogue pain scale (VAS) by using the scale in numbers from 0-10 cm in post anesthesia care unit.
  Note:
  Mild pain was considered score from 0 to 3, Moderate pain was labelled the score from 4 to 6 and Severe pain was considered the score from 7 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Dileep Kumar, FCPS, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: Yes
All IPD data will be shared through the publication but without the sharing the participants identities.
Supporting Information: SAP
Time Frame: After recruitment of sample size
Access Criteria: The data can be accessed by requesting the institutional ethical review committee and falling under the category of data sharing

REFERENCES:
- [Background] Ali MA, Shamim F, Chughtai S. Comparison between intravenous paracetamol and fentanyl for intraoperative and postoperative pain relief in dilatation and evacuation: Prospective, randomized interventional trial. J Anaesthesiol Clin Pharmacol. 2015 Jan-Mar;31(1):54-8. doi: 10.4103/0970-9185.150542. PMID 25788774